CLINICAL TRIAL: NCT06340061
Title: The Aim of This Study is to Investigate the Correlation Between the Severity of Glaucoma and Corneal Biomechanics as Well as Anterior Chamber Parameters.
Status: Active, not recruiting | Type: Observational
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Qianyu Wu
Record Dates: First submitted 2024-03-10; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group
  Interventions: Other: Observational study
- Control group

INTERVENTIONS:
Other: Observational study — The ocular biomechanical differences between the normal control group and primary glaucoma patients, including those treated with conventional medication, laser therapy, and surgery, were compared. Additionally, an investigation was conducted to explore the relationship between anterior chamber parameters, corneal biomechanics, and the severity of glaucoma
  Groups: Treatment group

SUMMARY:
The ocular biomechanical differences between the normal control group and primary glaucoma patients, including those treated with conventional medication, laser therapy, and surgery, were compared. Additionally, an investigation was conducted to explore the relationship between anterior chamber parameters, corneal biomechanics, and the severity of glaucoma

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of primary glaucoma.
* Must be able to cooperate to complete the inspection.

Exclusion Criteria:

* Secondary glaucoma.
* Corneal disease (E. g., keratitis, corneal scarring) that the investigator believes may affect the examination.
* trauma
* congenital eye malformations

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-10-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
IOP | through study completion, an average of 2 years.
  Intraocular pressure
bIOP | through study completion, an average of 2 years.
  Biomechanical intraocular pressure. Corneal Biomechanics Parameters.
ACD | through study completion, an average of 2 years.
  Anterior chamber depth. Anterior Chamber Parameters.
ACW | through study completion, an average of 2 years.
  Anterior chamber width. Anterior Chamber Parameters.
SSI | through study completion, an average of 2 years.
  Stress-strain index. Corneal Biomechanics Parameters.
VF | through study completion, an average of 2 years.
  visual field. The severity of glaucoma is mainly based on the damage of the visual field

CONTACTS AND LOCATIONS:
Overall Officials: Qian Liu, Principal Investigator — Henan Provincial People's Hospital, Henan Eye Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No